CLINICAL TRIAL: NCT03785795
Title: Optimizing and Validating an EMG-based Fetal Monitor to Identify True Preterm Labor
Brief Title: Multichannel EMG Diagnosing True Preterm Labor
Acronym: PTL
Status: Completed | Type: Observational
Sponsor: PreTeL, Inc (Industry)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: SBIR1.01
Record Dates: First submitted 2018-12-19; First posted 2018-12-24 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Pregnancy Preterm; Labor; Irregular; Preterm Labor
Keywords: Preterm labor detection; Labor detection; False labor
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Uncertain diagnosis of true labor: Patients who cannot be accurately classified as experiencing true labor or false labor based on standard clinical assessments.
  Interventions: Device: Uncertain diagnosis of true labor

INTERVENTIONS:
Device: Uncertain diagnosis of true labor — Multichannel EMG of uterine bioelectrical signals will be recorded using area sensors. The output of the synchronization calculations will be correlated with the time to delivery

SUMMARY:
We have designed new electromyography sensors for measuring uterine activity. These sensors are directional - they preferentially report uterine muscle contractions at specific locations, called regions. By measuring the synchronization of the regions of the uterus during contractions we intend to non-invasively determine if any patient is in-labor or not-in-labor. Accurately diagnosing true preterm labor allows timely intervention to avoid preterm birth; Accurately diagnosing false preterm labor avoids needlessly treating patients who would not benefit.

DETAILED DESCRIPTION:
The legacy device for assessing uterine contractions is the tocodynamometer (Toco). The Toco is plunger-driven device that measures the uterine shape change that occurs with a contraction. Toco only reports the timing of contractions, not the contraction strength, and cannot distinguish between false and true labor.

Our overarching goal is to validate our method of determining if a patient experiencing contractions is in true labor or false labor. We will accomplish this by applying new knowledge to an old technology - uterine EMG.

This trial is based on our advanced understanding of how the uterus generates coordinated contractions without a pacemaker or dedicated electrical conduction pathways - mechanotransduction and intrauterine pressure - but also uses bioelectrical signaling for local tissue recruitment.

The uterus emits bioelectrical signals with each contraction that can be detected by electromyography (EMG). To observe uterine bioelectrical signals, we created a novel EMG sensor, we call the "area sensor". This sensor is directional - capable of preferentially reporting muscle contractions from immediately below the sensor location.

In this clinical trial we use multiple area sensors placed on the maternal abdomen to directly observe how well the regional contractions are synchronized. Our hypothesis to be tested is that highly synchronized contractions predicts true labor, unsynchronized predicts false labor.

Patients with unclear labor status, or those in early labor will be studied. We will correlate the results of the synchronization analysis against the patient's progress over the ensuing 24 hours. These data will validate the ability to identify false and true labor using multichannel EMG and area sensors.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* One living fetus
* Experiencing frequent uterine contractions

Exclusion Criteria:

* Cervical dilation > 4 cm
* Ruptured membranes
* Maternal or fetal indications for immediate delivery

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Subjects must be pregnant
Study Population: Pregnant women with viable pregnancies who are experiencing uterine contractions will be studied. For each subject, her provider will not be certain if she is in true labor, or is experiencing false labor contractions. Other than experiencing contractions, subjects will have uncomplicated pregnancies. She will not have an indication for immediate delivery.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2018-11-25 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Validating prediction of true/false labor status with delivery within 24 hours | 24 hours
  The test device predicts delivery. The prediction on each subject will be compared against the observed delivery time.

SECONDARY OUTCOMES:
Establishing the range and trend of synchronized sensor readings | 48 hours
  The fraction of EMG channels active during each contraction, and the running average of the fraction, will be correlated with time to delivery

CONTACTS AND LOCATIONS:
Overall Officials: Roger C Young, MD, Principal Investigator — PreTeL, Inc
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Specific patient EMG tracings may be shared based on unique characteristics of pregnancy subsets.

REFERENCES:
- [Background] Young RC. Mechanotransduction mechanisms for coordinating uterine contractions in human labor. Reproduction. 2016 Aug;152(2):R51-61. doi: 10.1530/REP-16-0156. Epub 2016 May 10. PMID 27165050

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT03785795/Prot_SAP_000.pdf